CLINICAL TRIAL: NCT00997776
Title: Effect of Leg Strengthening Exercise After Hip Fracture
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcadia University (Other)
Responsible Party: Kathleen Kline Mangione, Professor, Arcadia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MANGIONE-LEG STRENGTH 2006; 1R03HD041944-01A1 (NIH)
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Hip Fractures
Keywords: Hip Fracture; Exercise; Rehabilitation; Functional Performance
MeSH Terms: conditions — Hip Fractures; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): High intensity lower extremity exercise
  Interventions: Other: progressive resistance exercise
- Attention control (Sham Comparator): lower extremity TENS
  Interventions: Other: TENS

INTERVENTIONS:
Other: progressive resistance exercise — lower extremity strengthening: 3 sets of 8 repetitions at the 8 repetition maximum (8RM)for the hip and knee extensors, hip abductors, plantarflexors twice weekly for 10 weeks.
  Other Names: strengthening exercise
  Arms: Exercise
Other: TENS — Transcutaneous electrical nerve stimulation (TENS) to elicit sensory information (comfortable tingling) for 7 minutes to bilateral muscle groups including the gluteal muscles, quadriceps, and gastroc-soleus muscles. TENS administered twice weekly for 10 weeks.
  Arms: Attention control

SUMMARY:
The purpose of this trial was to examine the effectiveness of a short-term leg strengthening exercise program compared to attention control on improving leg strength, walking speed and endurance, physical performance, and physical function one year after hip fracture.

DETAILED DESCRIPTION:
Poor functional outcomes are reported for the majority of older adults who sustain a hip fracture. The ability of hip fracture patients to make sustained functional improvements above and beyond natural recovery is unknown. It has been shown that gym-based programs can help old adults regain function after hip fracture. It is unclear if these results could be translated into the home setting that lacks the gym-based equipment, or if improvement would be sustainable. This program compares high intensity strength training performed in the home twice weekly for 10 weeks to an attention placebo control in which participants receive sensory electrical stimulation to leg muscles.

ELIGIBILITY:
Inclusion Criteria:

* Successful fixation (partial or total hip replacement or open reduction internal fixation) of a hip fracture within the last 6 months
* Were 65 years of age or older, were living at home prior to the fracture, had a physician referral and were discharged from physical therapy.

Exclusion Criteria:

* Medical history of unstable angina or uncompensated congestive heart failure, ongoing chemotherapy or renal dialysis, history of stroke with residual hemiplegia, Parkinson disease, absent sensation in the lower extremities due to sensory neuropathy, life expectancy of less than 6 months, and Folstein mental status scores < 20.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-08; Primary Completion 2006-01 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
lower extremity force production | one year after hip fracture

SECONDARY OUTCOMES:
six minute walk distance | one year post fracture
free and fast gait speed | one year post fracture
modified physical performance test | one year post fracture
SF-36 physical function | one year post fracture

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen K Mangione, PT, PhD, Principal Investigator — Arcadia University
Locations (1):
- Arcadia University, Glenside, Pennsylvania, United States